CLINICAL TRIAL: NCT03570346
Title: A Randomised, Double-Blind, Placebo Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics of Hemay005 in Healthy Subjects
Brief Title: Multiple Ascending Dose Study to Assess Safety and Pharmacokinetics of Hemay005 In Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Hemay Bio-Tech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM005PS1S03
Record Dates: First submitted 2018-06-17; First posted 2018-06-26 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemay005 (Experimental): 6 subjects in each cohort(15mg, 30mg, 60mg) will receive Hemay005
  Interventions: Drug: Hemay005
- Placebo (Placebo Comparator): 2 subjects in each cohort(15mg, 30mg, 60mg) will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hemay005 — Subjects will be randomized into 3 dose groups orally twice daily.
  Arms: Hemay005
Drug: Placebo — Subjects will be randomized into 3 dose groups orally twice daily.
  Arms: Placebo

SUMMARY:
Hemay005 is a novel phosphodiesterase type 4(PDE4) inhibitor being developed for the treatment of psoriasis. A total of approximately 24 subjects will be randomized into 3 cohorts(15mg, 30mg, 60mg), approximately 8 healthy subjects will be enrolled (6 active and 2 placebo) at each dose cohort. This study includes an 28-day Screening Period, a 1-day single dose and 7-days multiple doses Treatment Period, and an End of Study Visit occurring approximately 11days (±3 days) after study drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 to 60 years, male and female volunteers;
2. Male Bodyweight（BW）≥ 50kg, female Bodyweight（BW）≥ 45kg, Body mass index (BMI) in 18-28 (including upper and lower limit of the range);
3. All male subjects must agree and commit to the use of a reliable contraceptive regimen(including vasoligation, abstinence, using a condom) for the duration of the study(from screening until 6 months after the last dose), Female participants with a negative pregnancy test (serum) at both the screening visit and at Day-1, Female subjects and female partners of male subjects must agree and commit to the use of a reliable contraceptive regimen ( oral contraceptive medications or non-oral contraceptive medications) for the duration of the study(from screening until 6 months after the last dose);
4. Ability to understand and be willing to sign a written informed consent before study entry;
5. Subjects would have good communication with the investigator and could comply with protocol.

Exclusion Criteria:

1. A history of clinically severe gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, psychiatric disease or haematological disorders;
2. Have a known history of hypersensitivity to any medicine or food, or allergy to the test article or any of the excipient of the test article;
3. Have a gastrointestinal, hepatic or renal condition that may influence drug absorption or metabolism;
4. A history of chronic infection (ie, tuberculosis);
5. A medical history of any clinically significant medical disease or surgery within 4 weeks of the screening;
6. Clinically significant laboratory abnormal results at screening or prior to the first dose of study drug;
7. Clinically significant abnormal 12-lead ECG or vital signs ( systolic pressure <90 mmHg or >140 mmHg, diastolic pressure <50 mmHg or >90 mmHg; radial pulse rate <50 bpm or >100 bpm);
8. Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening;
9. Recent history of frequent alcohol consumption, defined by average intake of greater than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL of spirits with 40% alcohol content, or 150 mL wine), Participants who are unable to abstain from smoking during the study or quitting smoking for less than 3 months;
10. Positive urine screen for drug and cigarettes, positive breath test for alcohol;
11. Subjects who use soft drugs (ie marijuana )within 3 months of the screening and entire study duration or hard drugs (ie cocaine, phencyclidine ) within 1 year of the screening and entire study duration;
12. Dietary habits or food intolerances which will interfere with the requirements for participants to consume a standardised diet whilst confined to the clinical unit;
13. Participants who eat special food (Including grapefruit and/or Xanthine diet) for 14 days prior to dosing or any caffeine containing food or drinks, i.e. chocolate for 48 hours prior to dosing or drinking alcohol for 24 hours prior to dosing and not will stop to intake above food and drinks;
14. Use of any drug that inhibits or induces hepatic metabolism of drugs within 30 days of planned study drug administration and entire study duration (e.g. inducers: barbiturates, carbamazepine, rifampicin, phenytoin, glucocorticoid and omeprazole; inhibitors - Selective Serotonin Reuptake Inhibitors(SSRI )antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones and antihistamines);
15. Participant who received any medicine within 14 days of the initial dose of study drug;
16. Have received other clinical trials treatment within 3 months prior to study;
17. Participants who have donated of blood (>400 mL) within 4 weeks of the study, or plan to donate of blood during of the study and 4 weeks after the study;
18. Subjects cannot complete the study due to other reasons or by the investigator's judgment;
19. Pregnancy or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-10-20 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events. | Day1 up to Day20±3

SECONDARY OUTCOMES:
Cmax | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose on day 1 and day11
  Maximum observed plasma concentration
area under the curve from time zero to the last quantifiable concentration | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose on day 1 and day11
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration
area under the curve from time zero extrapolated to infinity | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose on day 1 and day11
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
t1/2 | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose on day 1 and day11
  Terminal elimination half-life
clearance CL/F | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose on day 1 and day11
  Apparent total plasma clearance
Vz/F | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose on day 1 and day11
  Apparent total volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Hongyun Wang, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided